CLINICAL TRIAL: NCT06332378
Title: Effect of Exercise Therapy on Type II Diabetic Neuropathic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Sobia Hasan (Other)
Responsible Party: Sponsor-Investigator, Dr. Sobia Hasan, Dr.Sobia Hasan, University of Karachi
Organization: University of Karachi (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sHasan
Record Dates: First submitted 2024-03-17; First posted 2024-03-27 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Nephropathy Type 2
Keywords: Exercise Therapy; Diabetic Neuropathies; Type 2 Diabetes Mellitus; Michigan Neuropathy Screening Instrument
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus, Type 2 | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ball training exercise (Experimental)
  Interventions: Other: Experimental group 1 :Ball training
- Frenkel training exercise (Experimental)
  Interventions: Other: Experimental group 2 :Frenkel Exercises
- control group (Other)
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Experimental group 1 :Ball training — Ball training Training in sitting position (the participants sat on the ball and did the exercises): holding balance position on the ball, active movements (flexion, extension, abduction, adduction) of one upper extremity, active movement of two upper extremities, trunk movements (bending forward and rotation), raising heel, raising toes, raising heel and toes simultaneously, resistance against perturbation, and weight shifting on ball and 2-Training in standing position: moving the ball up and down in a straight line with two upper extremities, moving the ball up and down in an oblique line with two upper extremities, moving the ball forward and backward with left and right lower extremities, moving the ball laterally with left and right lower extremities, throwing the ball against the wall with hand, throwing the ball against the wall with foot
  Arms: ball training exercise
Other: Experimental group 2 :Frenkel Exercises — Frenkel Exercises Supine position
  1. Flex and extend one leg, heel sliding down a straight line on table.
  2. Abduct and adduct leg with knee and hip extended, leg sliding on table. Sitting position
  1. Place foot on therapist's hand, which will change position. 2. Raise leg and put foot on traced footprint on the wall. 3. Rise and sit with knees together. Standing position
  1. Place foot forward and backward on a straight line.
  2. Walk along a winding strip.
  3. Walk between two parallel lines
  Arms: Frenkel training exercise
Other: Control Group — By using random allocation, the participants will divided into three groups: an intervention group (N=30) that receive ball training exercise, another intervention group (N=30) that receive Frenkel training exercise and a control group (N=30
  Arms: control group

SUMMARY:
The goal of this Randomized control trial (clinical trial) is to learn about the effect of Exercise therapy on Type II Diabetic Neuropathic Patient in Pakistan ,40-70 year's old patient, will be refer by physicians.

Exclusion criteria of the study will lower extremity complications such as fracture, having experience dislocation at least six months prior to the study, having any history of surgical operations in muscles, bones, and joints of lower extremities, suffering from musculoskeletal disorders such as rheumatoid arthritis and myopathy, middle ear and vestibular impairments (patients' self-report), knee joint flexion contracture, and interruption of the intervention sessions for more than two days..

The main question it aims to answer are:

1. To compare the effects of two therapeutic exercises on clinical balance measures on type II diabetic peripheral neuropathy patients.
2. Effectiveness of exercises using Swiss ball in lowering BMI.
3. To assess the effectiveness of exercise interventions on fasting blood sugar (FBS) levels and glycosylated hemoglobin (HbA1c) in individuals with Type II diabetes.
4. To evaluate the effectiveness of exercise interventions on autonomic nervous system activity in patients with Type II diabetic peripheral neuropathy.
5. To assess the comparative effectiveness of two therapeutic exercise interventions and a control group in improving the Michigan Neuropathy Screening Instrument (MNSI) score.

By using random allocation, the participants will divided into three groups: an intervention group (N=30) that receive ball training exercise, another intervention group (N=30) that receive Frenkel training exercise and a control group (N=30).

Each exercise session contain 5 min warm-up (stationary bike), 45 min exercise training (with 1 minute rest for every 5 minutes of exercise), and 5 min of cool down activities including stretching of the muscles involved in balance exercise (gluteal, erector spine, hamstring, rectus femorus, gastro soleus, and pectoral muscles). This make the participants' heart rate stable and prepare their muscles for optimal activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type II diabetic neuropathy
* 40-70 year's old patient, will be refer by physicians.

Exclusion Criteria:

* lower extremity complications fracture
* having experience dislocation at least six months prior to the study
* having any history of surgical operations in muscles, bones, and joints of lower extremities,
* suffering from musculoskeletal disorders such as rheumatoid arthritis and myopathy, middle ear and vestibular impairments (patients' self-report)
* knee joint flexion contracture
* interruption of the intervention sessions for more than two days

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
One Leg Stance | 6 weeks
  One Leg Stance assesses postural stability. This test includes standing on one foot without any help. This vary according to age.40-49 years-old (eyes open): 40 seconds. 50-59 years-old (eyes open): 37 seconds .
  60-69 years-old (eyes open): 26.9 seconds. 70-79 years-old (eyes open): 18.3 seconds. These are normal values less than normal values indicate postural instability
Berg Balance Scale | 6 weeks
  The Berg Balance Scale, is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete.
Timed Up and Go Test: | 6 weeks
  Measures the time it takes for an individual to stand up from a chair, walk three meters, turn around, walk back to the chair, and sit down. < 10 seconds = normal. < 20 seconds = good mobility; can walk outside alone; does not require a walking aid. < 30 seconds = walking and balance problems; cannot walk outside alone; requires walking aid.
Diabetic Neuropathy Symptom Score | 6 weeks
  Diabetic Neuropathy Symptom (DNS) score is a diabetic neuropathy screening consisting of scores from 1 to 4, and a score of ≥1 is considered significant. The severity of diabetic neuropathy was measured using an England score consisting of mild, moderate, and severe.
Hemoglobin A1C | 8 weeks
  HbA1c is short for glycated Haemoglobin. The test is also sometimes called Haemoglobin A1c. Haemoglobin (Hb) is the protein in red blood cells that carries oxygen through your body. HbA1c refers to glucose and haemoglobin joined together (the haemoglobin is 'glycated').An A1c level of 7 percent is considered high and means that 7% of the hemoglobin in your blood is saturated with sugar. HbA1c (%) levels of women and men in different age groups in HbA1c <6.5 and HbA1c ≥6.5 groups.
  1. 30-39: 5.34
  2. 40-49: 5.49
  3. 50-59 : 5.65. A1c levels of 6.5 or greater are considered diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Sobia Hasan, PhD*, Principal Investigator — Ameen Medical center; Aftab Ahmed Mirza Baig, PhD, Study Director — Iqra University, North Campus, Karachi, Pakistan
Locations (1):
- Ameen Medical & Dental Centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melese H, Alamer A, Hailu Temesgen M, Kahsay G. Effectiveness of Exercise Therapy on Gait Function in Diabetic Peripheral Neuropathy Patients: A Systematic Review of Randomized Controlled Trials. Diabetes Metab Syndr Obes. 2020 Aug 5;13:2753-2764. doi: 10.2147/DMSO.S261175. eCollection 2020. PMID 32848436
- [Background] Francia P, De Bellis A, Iannone G, Sinopoli R, Bocchi L, Anichini R. The Role of New Technological Opportunities and the Need to Evaluate the Activities Performed in the Prevention of Diabetic Foot with Exercise Therapy. Medicines (Basel). 2021 Dec 2;8(12):76. doi: 10.3390/medicines8120076. PMID 34940288